CLINICAL TRIAL: NCT01212913
Title: Comparison of a Basal Plus (Insulin Glargine/Insulin Glulisine) Regimen to Biphasic Insulin (InsulinAspart/Insulin Aspart Protamine 30/70) in T2DM Patients Who Require Insulin Intensification After Basal Insulin Optimization.
Brief Title: Comparison of Insulin Glargine/Insulin Glulisine Regimen to Insulin Aspart/Insulin Aspart Protamine 30/70 in Type 2 Diabetes Mellitus Patients (T2DM)
Acronym: B to B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04867; U1111-1117-2786 (Other: WHO)
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine; Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1: Basal plus (Experimental): Insulin glargine with dosage adjustment determined according to the mean value of the last three days Fasting Blood Glucose (FBG) Insulin glulisine, at initial dosing of 4IU, then weekly adjusted according to the mean value of the last three days PostPrandial Blood Glucose (PPBG)
  Interventions: Drug: INSULIN GLARGINE; Drug: INSULIN GLULISINE
- group 2: Biphasic insulin (Active Comparator): Insulin aspart/insulin aspart protamine 30/70 (novomix 30) given twice daily and titrated weekly (before breakfast and dinner) according to the lowest of three previous days' pre-meal levels (both breakfast and dinner). Target is 70 mg/dL < Pre-meal blood glucose (dinner and breakfast).
  Interventions: Drug: Insulin aspart

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution for injection Route of administration: subcutaneous Dose regimen: once daily
  Other Names: Lantus
  Arms: group 1: Basal plus
Drug: INSULIN GLULISINE — Pharmaceutical form: solution for injection Route of administration: subcutaneous Dose regimen: once daily
  Other Names: Apidra
  Arms: group 1: Basal plus
Drug: Insulin aspart — Pharmaceutical form: solution for injection Route of administration: subcutaneous Dose regimen: twice daily
  Other Names: NovoMix 30
  Arms: group 2: Biphasic insulin

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of hemoglobin A1c (HbA1c) control at six months between the basal plus one and the biphasic insulin regimen.

Secondary Objective:

To demonstrate favorable outcome for basal plus over biphasic insulin when it comes to comparing when both hemoglobin A1c (HbA1c) target goal achievement and non-hypoglycemic event is taken into account.

ELIGIBILITY:
Inclusion criteria:

1. Sub-optimally controlled Type 2 Diabetes Mellitus (T2DM) patients treated with insulin glargine for a minimum of 3 months:

   * Sub-optimal: HbA1c level >7% and fasting blood glucose <130mg/dL
2. Male or Female ≥18 years old
3. Body Mass Index (BMI) <40
4. 10% ≥HbA1c ≥7%
5. If taking Oral anti-diabetics (OADs), must be on stable dose for at least 1 months
6. Patients willing to sign data release consent form

Exclusion criteria:

1. Diabetes other than T2DM
2. Enrolled in other clinical trials
3. Previous treatment with an insulin other than insulin glargine
4. Treatment with Glucagon-like peptide-1 (GLP-1) receptor agonists or with Di Peptidyl Peptidase 4 (DPP-IV) inhibitors
5. Pregnant or lactating women
6. Contraindicated to Lantus (insulin glargine) / Apidra (insulin glulisine) / Novomix 30 (insulin aspart)
7. Treatment with systemic corticoid steroids within the last 3 months prior to study enter
8. Treatment with any investigational product within the last 3 months prior to study entry

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c level (HbA1c) | At 6 months of treatment

SECONDARY OUTCOMES:
Rate of hypoglycemic events (total, severe, nocturnal) | from baseline to the study endpoint (over 6 months of treatment)
Proportion of patients with HbA1c < 7% | from baseline to the study endpoint (over 6 months of treatment)
Change in body weight | from baseline to the study endpoint (over 6 months of treatment)
Reactive Oxidative Stress (ROS) level changes | from baseline to the study endpoint (over 6 months of treatment)
Change in Quality of Life | from baseline to the study endpoint (over 6 months of treatment)
Continuous Glucose Monitoring System (CGMS) data | at baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Administrative Office, Seoul, South Korea

REFERENCES:
- [Derived] Jin SM, Kim JH, Min KW, Lee JH, Ahn KJ, Park JH, Jang HC, Park SW, Lee KW, Won KC, Kim YI, Chung CH, Park TS, Lee JH, Lee MK. Basal-prandial versus premixed insulin in patients with type 2 diabetes requiring insulin intensification after basal insulin optimization: A 24-week randomized non-inferiority trial. J Diabetes. 2016 May;8(3):405-13. doi: 10.1111/1753-0407.12312. Epub 2015 Jun 29. PMID 25952532